CLINICAL TRIAL: NCT02830698
Title: Abdominal Pain Disorders Functional in Children: Impact of Hypno-analgesia on the Autonomic Balance. A Prospective Single-center Study
Brief Title: Abdominal Pain Disorders Functional in Children: Impact of Hypno-analgesia on the Autonomic Balance
Status: Terminated | Type: Observational
Why Stopped: Recruitment difficulties.
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1608081; 2016-A00868-43 (Other: ANSM)
Record Dates: First submitted 2016-06-21; First posted 2016-07-13 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Child; Abdominal Pain
Keywords: Nervous System; Hypnosis; Electrocardiography, Ambulatory; Abdominal pain disorders functional
MeSH Terms: conditions — Abdominal Pain; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Abdominal pain disorders functional (including functional dyspepsia, irritable bowel syndrome, abdominal migraine, functional abdominal pain) is a very common disease in the pediatric population, where classical medical treatment does not always prove effective. This clinical entity has an impact on the individual physiological balance particularly on the autonomic regulation. Studies concerning adults with irritable bowel syndrome, showed significant changes in heart rate variability indices (HRV: heart rate variability).

The study of time and frequency domain analysis of HRV allows noninvasive and reproducible assessment of the cardiac sympathetic and parasympathetic tone.

The investigators hypothesize that the sympathovagal balance could be altered in children in case of prolonged nociceptive stress as the investigators find it especially in irritable bowel syndrome and functional abdominal pain. In recent years, the control of pediatric pain experienced considerable growth through hypnosis techniques and several studies have shown analgesic efficacy with a beneficial effect in terms of quality of life in children.

Our study aims to assess the impact of the hypno-analgesia treatment of Abdominal pain disorders functional on sympathovagal balance. The investigators propose to realize in 7 to 18 years old children with Abdominal pain disorders functional a single center prospective study to highlight after a standardized hypnosis program, changes in the time and frequency domain indices of heart rate variability and clinical or quality of life parameters. The primary endpoint will be the high frequency HF indice. Secondary endpoints will be the other indices of HRV (Ptot, VLF, LF, ratio LF / HF, SDNN, SDANN, pNN50, RMSSD), the Quality of Life Questionnaire values (PedsQL ™ 4.0) a pain scale and the composite score of Francis.

ELIGIBILITY:
Inclusion Criteria:

* Parents affiliates or entitled to a social security scheme
* Consent form signed by the holder of parental authority

Exclusion Criteria:

* Child with pathologies reaching the central nervous system or the brain stem.
* Children with a severe pathology of cardio-respiratory or heart being referred to treatment.
* Children requiring emergency surgery or trauma or septic or inflammatory context.
* Children with psychiatric disorders or mental retardation proven.
* Children who have already used the earlier hypnosis.
* Children not speaking French language.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Indices of autonomic nervous system in a pediatric population with Abdominal pain disorders functional
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
high frequency | One month after the hypno-analgesic therapeutic program
  measured with the holter

SECONDARY OUTCOMES:
composite score of Francis | One month after the hypno-analgesic therapeutic program
  severity scale of syndrome (pain intensity)
Pediatric Quality of Life inventory | One month after the hypno-analgesic therapeutic program
a chronic abdominal pain scale | One month after the hypno-analgesic therapeutic program
  adaptation of Francis composite scale for chronic abdominal pain
a severity of functional dyspepsia scale | One month after the hypno-analgesic therapeutic program
  adaptation of Francis composite scale for functional dyspepsia
a severity of abdominal migraine scale | One month after the hypno-analgesic therapeutic program
  adaptation of Francis composite scale for abdominal migraine
SDNN (standard deviation of all NN intervals) | One month after the hypno-analgesic therapeutic program
  measured with the holter
SDANN (standard deviation of the averages of NN intervals in all 5 min segments of the entire recording) | One month after the hypno-analgesic therapeutic program
  measured with the holter
RMSSD (the square root of the mean of the sum of the squares of difference between adjacent NN intervals) | One month after the hypno-analgesic therapeutic program
  measured with the holter
pNN50 (the number of pairs of adjacent NN intervals differing by more than 50 ms dived by the total number of all NN intervals) | One month after the hypno-analgesic therapeutic program
  measured with the holter
TP (total power) | One month after the hypno-analgesic therapeutic program
  measured with the holter
VLF (very low frequency component) | One month after the hypno-analgesic therapeutic program
  measured with the holter
LF (low frequency component) | One month after the hypno-analgesic therapeutic program
  measured with the holter
ratio LF/ HF | One month after the hypno-analgesic therapeutic program
  measured with the holter

CONTACTS AND LOCATIONS:
Overall Officials: Hugues PATURAL, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- Centre Hospitalier Universitaire de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No